CLINICAL TRIAL: NCT01410045
Title: Cryopreservation of Ovarian Cortex in Girls With Turner Syndrome : Karyotypic, Clinical and Hormonal Criteria to Screen Patients
Brief Title: Cryopreservation of Ovarian Cortex in Girls With Turner Syndrome
Acronym: CRYO-X0
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P081204
Record Dates: First submitted 2011-06-28; First posted 2011-08-04 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Turner Syndrome; Ovarian Insufficiency
Keywords: Turner syndrome; infertility; ovarian insufficiency; ovarian cryopreservation
MeSH Terms: conditions — Turner Syndrome; Infertility | interventions — Ovariectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): Ovariectomy
  Interventions: Procedure: Ovariectomy

INTERVENTIONS:
Procedure: Ovariectomy — Ovarian cryopreservation has been used in an effort to preserve fertility in patients undergoing treatments which lead to premature and severe ovarian insufficiency.

SUMMARY:
Ovarian insufficiency is common in Turner syndrome related to premature and rapid follicular apoptosis and spontaneous pregnancies are rare in this population. Ovarian cryopreservation has been used in an effort to preserve fertility in patients undergoing treatments which lead to premature and severe ovarian insufficiency. This study aims to assess the relevance of ovarian tissue cryopreservation in girls with Turner syndrome. Based on ovarian follicular density as primary outcome and karyotypic, clinical and hormonal markers as secondary outcomes, analysis of the study will allow to select the patients to whom the procedure would benefit the most.

DETAILED DESCRIPTION:
Turner syndrome (TS) is characterized by the absence of all or part of a normal second X chromosome and occurs in about 1/2,500 live-born girls. Spontaneous fertility is rare among patients with TS related to premature apoptosis of ovarian follicles. Spontaneous puberty and fertility has been reported mostly in patients with mosaic karyotype or small X deletions.

There is robust evidence that follicles can be observed in ovaries in girls with TS. However, follicular density and quality seems to be largely influenced by karyotype, ovarian morphology and endocrine competence. There are no clear-cut clinical or hormonal markers to assess the ovarian reserve in girls with TS but markers of ovarian function used in women with premature ovarian insufficiency are measured. In TS, it is now fundamental to be able to evaluate the prognosis of the ovarian function and the degree of fertility to provide the relevant information to girls and their parents and to discuss possibilities of motherhood if any.

Ovarian cryopreservation has been used in an effort to preserve fertility in patients undergoing treatments which lead to premature and severe ovarian insufficiency. This study aims to assess the relevance of ovarian tissue cryopreservation in girls with Turner syndrome. Based on ovarian follicular density as primary outcome and karyotypic, clinical and hormonal markers as secondary outcomes, analysis of the study will allow to screen the patients to whom the procedure would benefit the most.

Girls who will be operated will accept to come for a follow-up visit at one and 12 months after the surgery. It is expected to have clinical and hormonal information through a long follow up performed by the referred paediatrician.

Results of the study will allow us to select patients with TS who will benefit the most of this fertility preservation procedure based on karyotypic, clinical and hormonal profile.

ELIGIBILITY:
Inclusion criteria :

* girls aged from 1 to 25 years included,
* with Turner syndrome or mosaic
* patients aged more than 18 will only have ovarian insufficiency dated less than 5 years
* without any severe disease, particularly of cardiovascular type
* whose agreement to participate to the study has been signed by the parents
* whose agreement to participate to the study has been signed by majority age patient

Exclusion criteria :

* girls aged less than one year and over 25 years old
* if any surgery would be contra-indicated
* ovary alone presence
* Well-known infection by HIV, and/or HBV, and/or HCV and/or syphilis TPHA VDRL
* No social coverage affiliate

Ages: 1 Year to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01-16 (Actual); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
the ovarian follicular density | at the time of the ovariectomy
  the specific measure is the ovarian follicular density which will allow to Identify criteria, to predict existence or absence of ovarian follicles at the time of the surgery

SECONDARY OUTCOMES:
measure hormonal markers | Before the ovariectomy, 1 month and 12 months after the ovariectomy
  measure hormonal markers as FSH, AMH, Inhibine B and estradiol before, at one month and one year after the ovariectomy

CONTACTS AND LOCATIONS:
Overall Officials: Lise Duranteau, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No